CLINICAL TRIAL: NCT01115634
Title: Autologous Transplantation of Cultured Fibroblast for Facial Contour Deformities
Brief Title: Autologous Fibroblast Transplantation in Facial Deformities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-skin-002
Record Dates: First submitted 2010-05-01; First posted 2010-05-04 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2010-05

CONDITIONS: Nasolabial Folds; Glabellar Crease; Deep Wrinkles of the Forehead; Acne Scars
Keywords: Fibroblast; Cell transplantation; Facial deformities
MeSH Terms: interventions — Carboxylesterase; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fibroblast (Experimental): Injection of autologous cultured fibroblast
  Interventions: Biological: Fibroblast; Biological: fibroblast and gel

INTERVENTIONS:
Biological: Fibroblast — 20 million cell in three injection
  Other Names: cell alone
Biological: fibroblast and gel — 20 million cell in three injection plus filler

SUMMARY:
Beautiful skin requires maintenance of proper care. Skin exercise, protections from direct sunlight or harsh wind, and maintaining a healthy diet are some of the ways of having a good and radiant skin. However despite all the care taken passage of time will bring about conditions that will automatically lead to skin aging, which may require certain therapeutic, care. Fibroblasts are cells that synthesize the extracellular matrix and collagen and play a critical role in wound healing and maintenance of healthy skin. Loosing of fibroblast cell is the main problem in aging and wrinkles and non-healed skin wounds. Therefore proliferation of skin fibroblast along with differentiation of stem cells in the skin tissue is the best method for healing.

DETAILED DESCRIPTION:
Autologous cultured fibroblast is derived from in vitro expansion of fibroblasts harvested from the patient's normal skin. Biopsies from behind a patient's ear are the source of fibroblasts, which are isolated, expanded through cell culture, and used for the correction of facial contour deformities such as nasolabial folds, glabellar crease, deep wrinkles of the forehead, and acne scars. Prior to final packaging, cell viability is assessed to be at least 85%.

Each single use container of autologous cultured fibroblasts has approximately 20 million cells aseptically processed and suspended in 1 mL of sterile, buffered Dulbecco's Modified Eagles Medium (DMEM). Both the biopsy transport media and the cell culture media contain gentamicin. Residual quantities of gentamicin up to 5 µg/mL may be present in the Cell product

ELIGIBILITY:
Inclusion Criteria:

* Available and willing to attend all follow-up visits.
* Age > 18 years.
* Able and willing to give informed consent.

Exclusion Criteria:

* Known allergy or sensitivity to collagen fillers
* The subject has received a soft tissue augmentation to the area to be treated within the last 6 months.
* Subject is unwilling to forgo any cosmetic augmentation procedures for the duration of the study.
* The subject has received autologous fat transfer in the last 6 months.
* Subject is suffering from facial Kaposi's sarcoma.
* The subject has active skin diseases or inflammation on or near the area of injection
* positive HIV, HBV, HCV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
2-point shift in at least one treated area using a standardized 7-point photoguide | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Shafiyan, MD, Principal Investigator — Royan Institute; Nasser Aghdami, MD., PhD, Study Director — Royan Institute
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Salehi Z, Shams-Ghahfarokhi M, Razzaghi-Abyaneh M. Internal Transcribed Spacer rDNA and TEF-1alpha Gene Sequencing of Pathogenic Dermatophyte Species and Differentiation of Closely Related Species Using PCR-RFLP of The Topoisomerase II. Cell J. 2020 Apr;22(1):85-91. doi: 10.22074/cellj.2020.6372. Epub 2019 Sep 8. PMID 31606971
- [Derived] Bajouri A, Orouji Z, Taghiabadi E, Nazari A, Shahbazi A, Fallah N, Mohammadi P, Rezvani M, Jouyandeh Z, Vaezirad F, Khalajasadi Z, Ghasemi M, Fanni A, Haji Hosseinali S, Alizadeh A, Baharvand H, Shafieyan S, Aghdami N. Long-Term Follow-up of Autologous Fibroblast Transplantation for Facial Contour Deformities, A Non-Randomized Phase IIa Clinical Trial. Cell J. 2020 Apr;22(1):75-84. doi: 10.22074/cellj.2020.6340. Epub 2019 Sep 8. PMID 31606970
- See also: Related Info — http://www.royaninstitute.org